CLINICAL TRIAL: NCT04382079
Title: Effects of Honey and Propolis on Head and Neck Cancer Patients With Oral Mucositis: a Randomized Controlled Trial
Brief Title: Honey Products for Cancer Patients With Oral Mucositis: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N202001041
Record Dates: First submitted 2020-05-03; First posted 2020-05-11 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2020-04

CONDITIONS: Oral Mucositis
Keywords: head and neck cancer; mucositis; honey; Taiwanese green propolis; intelligent care
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Mucositis | interventions — Honey; Propolis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- honey (Experimental): Honey, 10 grams per pack, calories 33.4 calories, protein 0.05 grams, fat 0.07 grams, fructose + glucose 7.0 grams, sodium 0 mg.
  Usage is three times a day after three meals. After oral care is required before use, use 10 grams of longan honey, circulate in the oral cavity for at least 30 seconds, and slowly swallow. Do not eat, drink, or gargle within 30 minutes of use.
  Interventions: Dietary Supplement: honey
- propolis (Experimental): Oil-soluble green propolis, propolis 100 mg / mL, dilute green propolis 200 times with edible oil, drink 0.5 mL each time, 3 times a day (a total of 50 mg).
  Usage: three times a day, after three meals. After oral care is required before use, draw about 0.5ml of green propolis into the mouth, circulate in the oral cavity for at least 30 seconds, and slowly swallow. Do not eat, drink or gargle within 30 minutes of use.
  Interventions: Dietary Supplement: propolis
- control (No Intervention): Routine care to encourage oral care three times a day.

INTERVENTIONS:
Dietary Supplement: honey — Since the patient received radiation therapy, Taiwan Longan Honey has been used for a total of eight weeks.
  Understand the changes of oral mucositis and various symptoms during this period
  Arms: honey
Dietary Supplement: propolis — Since the patient received radiation therapy, Taiwan green propolis has been used for a total of eight weeks.
  Understand the changes of oral mucositis and various symptoms during this period
  Arms: propolis

SUMMARY:
The investigators plan to conduct a 3-year pioneering care research project for mucositis in cancer patients. These include: (1) an analysis of the incidence and severity of mucositis, severity, treatment methods, and treatment costs; (2) an RCT comparing the effectiveness of honey, Taiwan green propolis, and usual care in mucositis of cancer patients; (3) monitoring of related symptom changes using a smart bracelet device; (4) a measurement of IL-1, IL-6, IL-10, and TNF in saliva and (4) modeling of the trend of mucositis for alertness and search of essential parameters of the complications.

DETAILED DESCRIPTION:
Mucositis is common among cancer patients receiving radiotherapy and chemotherapy. A total of 80-100% of the patients are suffering from the mucositis pain; their regular dieting is disturbed, nutritional status deteriorated, and even treatment discontinued. Some self-paid medications like glutamine have been used to prevent mucositis before and during radiotherapy/chemotherapy. However, the cost of glutamine is relatively high (NT15,000 month/person) and its treatment efficacy and side effects are still to be determined. Randomized controlled trials (RCTs) and experiments have shown that honey and propolis may be used for the management of mucositis. Taiwan is a country of rich agriculture with unique bee products among which the longan honey demonstrates the most significant antibacterial effects; the green propolis has also been proved to comprise antibacterial, anti-inflammatory, and antioxidant effects. However, none of these propolis products have been specifically trialed for the management of mucositis of cancer patients.

Bee products have been concerned as potential sources of natural antioxidants such as flavonoids, phenolic acids, and terpenoids. Their potential treatment effects have caught the attention of the medical community. Accumulating evidence is supporting the use of bee products in mucositis caused by chemotherapy, radiotherapy, or both. However, systematic review and meta-analysis have suggested a low quality of the included RCTs, and this affects the applicability of the evidence in the real clinical scenario.

The investigators plan to conduct a 3-year pioneering care research project for mucositis in cancer patients. These include: (1) an analysis of the incidence and severity of mucositis, severity, treatment methods, and treatment costs; (2) an RCT comparing the effectiveness of honey, Taiwan green propolis, and usual care in mucositis of cancer patients; (3) monitoring of related symptom changes using a smart bracelet device; (4) a measurement of IL-1, IL-6, IL-10, and TNF in saliva and (4) modeling of the trend of mucositis for alertness and search of essential parameters of the complications. In the first year, our project will focus on the analysis of the incidence and severity of mucositis, treatment methods, and treatment costs. In the second year, the planned RCT will be carried out and changes in heart rate, stress, and fatigue of the patients are to be collected using the smart bracelet. In the third year, the investigators will conduct a deep machine learning of the clinical and serial test data to predict the changes in symptoms. The modeling is anticipated to provide important parameter combinations that assist the alerting of possible severe complications. The overall findings of this project shall the strategical references for applying bee products in the prevention and treatment of mucositis in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age≧20 years old
* diagnosed as head and neck cancer patients
* Plan to Receive radiation therapy
* Consciousness, ability to complete research assessment and willing to participate in research
* Patients can be communicated in Mandarin and Taiwanese, and complete the questionnaire on their own or with the help of researchers.

Exclusion Criteria:

* History of allergic to honey, propolis, various pollen, alcohol
* People with mental disorders or cognitive dysfunction
* Diabetes mellitus
* Critical of end of life patient

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
oral mucositis | twelve weeks
  measurement tool: National Cancer Institute Common Terminology Criteria for Adverse Events and The World Health Organization grading system

SECONDARY OUTCOMES:
Numerical Rating Scale | twelve weeks
  measurement tool:Numerical Rating Scale,for pain status, range from 0 to 10, 10 was the most pain, 0 was no pain.
Xerostomia | twelve weeks
  measurement tool: Xerostomia Questionnaire
Functional Assessment of Cancer Therapy Scale- Head and Neck | twelve weeks
  measurement tool : Functional Assessment of Cancer Therapy Scale- Head and Neck, for patient's Quality of life (QoL), range from 0 to 100, score 100 means better outcome.
fatigue--Brief-Fatigue Inventory | Brief-Fatigue Inventory for two weeks.
  measurement tool: Brief-Fatigue Inventory, range 0 to 10, 10 was the worst fatigue.
fatigue--Visual Analogue Scale | Visual Analogue Scale for fatigue for twelve weeks.
  measurement tool: Visual Analogue Scale for fatigue, range 0 to 10, 10 was the worst fatigue.
IL-1, IL-6, IL-10,TNF | radiotherapy on Day 0, on the 7th, 14th, 21st day and on an average of 28 st day.
  The patient collected this saliva before the start of radiotherapy, on the 7th, 14th, 21st day and at the end of radiation therapy, a total of 5 tubes of saliva at a time

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Wei Huang, PhD, Study Chair — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
oral mucositis severity, fatigue, pain, quality of life
Supporting Information: Study Protocol, CSR
Time Frame: Before radiotherapy, until 12 weeks later
Access Criteria: Professor Huang will review the application to share IPD.

REFERENCES:
- [Derived] Jen SC, Chen YW, Tsai JT, Kuo CC, Ting LL, Huang WY, Huang TW, Chen JH, Gautama MSN. Effects of honey and Taiwanese green propolis on oral mucositis and quality of life in head and neck cancer patients undergoing radiotherapy: a randomized controlled trial. Food Funct. 2025 Jun 16;16(12):4958-4969. doi: 10.1039/d5fo00067j. PMID 40424080